CLINICAL TRIAL: NCT00260650
Title: Heart PACT: Patient Activation in High-Risk Patients With Heart Failure
Brief Title: Patient Activation in High-Risk Patients With Heart Failure
Acronym: HeartPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NRI 04-252
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
Keywords: heart failure, congestive; self-care; quality of life; health behavior
MeSH Terms: conditions — Heart Failure; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart PACT Program (Experimental): Heart PACT Program - patient activation intervention
  Interventions: Behavioral: Heart PACT Program
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Heart PACT Program — patient activation intervention
  Arms: Heart PACT Program

SUMMARY:
The purpose of this study was to determine the efficacy of a self-management program, called the Heart PACT Program, compared to usual health care in patients with heart failure. Outcomes measured were patient activation (skills needed to maintain function, collaborate with providers, and access care), self-care management, hospitalizations and emergency department visits.

DETAILED DESCRIPTION:
Background:

Heart failure (HF) places an enormous burden on patients, their families, health care systems and society. Readmission for HF occurs within 30 days following 20 percent of discharges from the VA system with similar rates in the Medicare health care system. Few studies have examined whether chronic heart failure (HF) outcomes can be improved by increasing patient engagement (known as activation) in care and capabilities for self-care management.

Objectives:

The objective was to determine the efficacy of a patient activation (Heart PACT) intervention compared to usual care on activation, self-care management, hospitalizations and emergency room visits in patients with HF.

Methods:

This study employed a randomized, 2-group, repeated-measures design at a single VA site. Following consent, 84 participants were stratified by activation level and randomly assigned to usual care (n = 41), or usual care plus the Heart PACT intervention (n = 43). The primary outcomes and measures were patient activation using the Patient Activation Measure (PAM); self-management using the Self-Care of Heart Failure Index (SCHFI) and the Medical Outcomes Study (MOS) Specific Adherence Scale; and hospitalizations and emergency room visits using self-report and VA databases. The Heart PACT intervention consisted of individual meetings and phone contacts over 6 months. The intervention leaders collaborated with patients to increase activation and improve HF self-management behaviors, such as adhering to medications and implementing health behavior goals. The primary analyses were 2 (group: control vs. intervention) x 3 (time) repeated measures analyses of variance.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

This study was done at the VA San Diego Healthcare System only. Participants must live in San Diego and meet all of the following inclusion criteria:

* Has VA primary care provider for heart failure care
* Hospitalization or emergency department visit for treatment of HF within past 12 months. Hospital discharge must be at least one month prior to study enrollment.

Hospitalization diagnoses may include: acute myocardial infarction (MI) or acute coronary syndrome with LV dysfunction (EF <40%); status post coronary bypass graft surgery with LV dysfunction (EF < 40%)

* Documented heart failure (systolic or diastolic dysfunction) by echocardiogram or physician diagnosis and Stage C heart failure
* 18 years of age or older
* Read and speak English
* Have telephone access

Exclusion Criteria:

Patients will be excluded if they meet any of these criteria:

* Are unable to give written informed consent
* Have had a major acute medical problem (e.g., stroke, acute MI, CABG, or percutaneous intervention), or are considered medically unstable within the prior month
* Have a history of severe pulmonary disease, renal disease requiring dialysis, severe hepatic disease, severe aortic or mitral stenosis, constrictive pericarditis, or cardiac transplant
* Have a left ventricular assist device (LVAD)
* Have a bi-ventricular pacemaker or implantable cardioverter defibrillator (ICD) placement in the past 1 month
* Have a life expectancy of less than 1 year
* Have current acute psychiatric problems, active substance abuse or homelessness
* Are participating in an ongoing clinical drug trial.
* Enrolled in specialty HF care via the HF Program or telehealth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
patient activation | baseline, 3 months, 6 months

SECONDARY OUTCOMES:
self-management | baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Gardetto, PhD NP, Principal Investigator — VASDHS
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Background] Riegel B, Moser DK, Rayens MK, Carlson B, Pressler SJ, Shively M, Albert NM, Armola RR, Evangelista L, Westlake C, Sethares K; Heart Failure Trialists Collaborators. Ethnic differences in quality of life in persons with heart failure. J Card Fail. 2008 Feb;14(1):41-7. doi: 10.1016/j.cardfail.2007.09.008. PMID 18226772
- [Background] McKibbin CL, Shively M, Glaser D, Kodiath M, Kelly A, Bormann JE, Stepnowsky C, Smith T. Readiness to change in heart failure patients: Adaptation of a pain readiness to change measure. Clinical Gerontologist. 2007 Oct 1; 31(2):33-43.